CLINICAL TRIAL: NCT06315738
Title: Randomized, Controlled, Phase 1-2 Open Label Study of ST266 IV Administration to Assess the Safety, Tolerability, and Preliminary Efficacy of ST266 in Infants With Necrotizing Enterocolitis
Brief Title: Study to Assess the Safety, Tolerability, and Preliminary Efficacy of ST266 in Infants With Necrotizing Enterocolitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST266-NEC-201
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing Enterocolitis; NEC
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - lower dose active + SOC treatment vs. SOC alone in higher weight range (Other): Infants with weight at diagnosis of NEC ≥1000 g and ≤3000 g; 0.5 mL/kg of ST266, QD, + Standard of Care (SOC) treatment (n=6); SOC (n=3)
  Interventions: Biological: ST266
- Cohort 2 - higher dose active + SOC treatment vs. SOC alone in higher weight range (Other): Infants with weight at diagnosis of NEC ≥1000 g and ≤3000 g; 1.0 mL/kg of ST266, QD; + Standard of Care (SOC) treatment (n=6); SOC (n=3)
  Interventions: Biological: ST266
- Cohort 3 - lower dose active + SOC treatment vs. SOC alone in lower weight range (Other): Infants with weight at diagnosis of NEC ≥800 g and ≤999 g; 0.5 mL/kg of ST266, QD; + Standard of Care (SOC) treatment (n=6); SOC (n=3)
  Interventions: Biological: ST266
- Cohort 4 - higher dose active + SOC treatment vs. SOC alone in lower weight range (Other): Infants with weight at diagnosis of NEC ≥800 g and ≤999 g; 1.0 mL/kg of ST266, QD; + Standard of Care (SOC) treatment (n=6); SOC (n=3)
  Interventions: Biological: ST266

INTERVENTIONS:
Biological: ST266 — Patients randomized to investigative drug product (ST266) will receive either 0.5 mL/kg or 1.0 mL/kg of ST266 QD in addition to Standard of Care treatment; Patients randomized to SOC will receive standard of care treatment only.

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of two dose levels (0.5 mL/kg and 1.0 mL/kg) of once daily (QD) via IV route of administration of ST266 in treating patients with Bell's stage IIA or higher medical NEC by incidence of treatment emergent adverse events (TEAEs) and SAEs, with a secondary objective to assess preliminary efficacy of the same two dose levels (0.5 mL/kg and 1.0 mL/kg) of QD via IV route of administration of ST266 in treating patients with Bell's stage IIA or higher medical NEC.

DETAILED DESCRIPTION:
This Phase 1-2 clinical trial is a randomized, controlled, open-label study using a sequential cohort design. Assignment to cohorts will be based on the following dosages and weight ranges: 0.5 mL/kg and 1.0 mL/kg; weight ≥1000 g and ≤3000 g, and weight ≥800 g and ≤999 g.

In each cohort, patients will be randomized to either ST266 + SOC or SOC alone. The first 3 patients randomized to ST266 will be staggered, where each patient must complete their 10 day treatment cycle and 1 month follow up visit and be evaluated by the Data Safety Monitoring Board (DSMB), before dosing of the next patient occurs. Patients randomized to SOC alone will follow the treatment plan as dictated by the Investigator or licensed medical designee and will be evaluated for the same inclusion/exclusion criteria and selected endpoints for analysis. If for any reason a patient is withdrawn, the decision for replacement will be determined by the DSMB.

Dosing for the next cohort will occur after review of safety data up to and including Day 28/1 Month from all patients in the previous cohort. The DSMB reviews will include comprehensive safety data analysis of data available at that time.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born from ≥26 weeks gestational age to 40 weeks gestational age; up to 40 weeks postmenstrual gestational age (gestational age plus chronological age in terms of weeks) with current weight at diagnosis of NEC between ≥800g and ≤3000g as a result of prematurity and/or IUGR. Parent(s)/legal medical representative(s) voluntarily provides written consent prior to study enrollment.
2. Minimum Bell stage IIA NEC diagnosis by radiologic confirmed pneumatosis intestinalis and may include intestinal dilation and ileus.

Exclusion Criteria:

1. Infants with abdominal perforation at less than 10 days of life
2. Not expected to survive ≥2 weeks or born with a lethal condition requiring hospice or palliative care (e.g., disease has progressed to NEC totalis, or patient has multi-organ system failure).
3. Born with major congenital anomalies such as cardiac defects (e.g., Tetralogy of Fallot) or chromosomal disorders/anomalies (e.g., neural tube defect).
4. Mother's receipt of any investigational product during pregnancy.
5. Infants with malignancies (e.g., neoplastic cell growth as a solid tumor or a blood neoplasm, such as congenital leukemia).
6. Infants with hypercoagulability disorders (any active thrombosis, diagnosis of disseminated intravascular coagulation or other acquired/inherited disorders (i.e., hemophilia) of coagulation.
7. Infants with a known immunodeficiency (such as galactosemia or agranulocytosis).
8. Infants with anatomic defects that require surgical intervention.
9. Infants with persistent pulmonary hypertension of newborn.
10. Infants with any congenital or acquired gastrointestinal pathology that preclude feeds within 7 days after birth (e.g., duodenal atresia).
11. Infants who have hypoxic ischemic injury (perinatal asphyxia).
12. Infants with polycythemia (at time of treatment) (>22 g/dL).
13. Positive maternal human immunodeficiency virus status.
14. History of maternal drug abuse (such as amphetamines, opiates, cocaine). This does not include marijuana, or prescription medications for treatment of drug abuse.
15. Considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
16. Infants diagnosed with NEC who will require immediate surgical intervention.

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability endpoint: incidence of adverse events | From date of randomization through 24 months of age
  Patients will be assessed for safety and tolerability of ST266 treatment given IV (two dose options: 0.5mL/kg or 1.0mL/kg) via review of treatment emergent adverse events (TEAEs). AEs are defined as per the International Neonatal Consortium (INC) neonatal AE severity scale (NAESS): Mild, Moderate, Severe, Life Threatening, Death. Relatedness to study drug (ST266) will also be assessed.
Safety and Tolerability endpoint: incidence of serious adverse events | From date of randomization through 24 months of age
  Patients will be assessed for safety and tolerability of ST266 treatment given IV (two dose options: 0.5mL/kg or 1.0mL/kg) via review of serious adverse events, defined as: any event that results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or may jeopardize patient so that requires intervention to prevent prior noted outcomes (includes study drug related dose-limiting toxicities and infusion reactions)
Safety and Tolerability endpoint: Changes in labs and vitals relative to disease progression | From date of randomization through 24 months of age
  Patients will be assessed for safety and tolerability of ST266 treatment given IV (two dose options: 0.5mL/kg or 1.0mL/kg) by evaluating clinically significant changes in labs and vitals as to relatedness to disease progression and study drug effects, including assessment of vital signs (temperature, systolic and Mean arterial blood pressure (mmHg), respiratory rate, heart rate, and percent oxygen saturation as measured by pulse oximetry as noted in The Harriet Lane Handbook, 21st ed., 2018), and hematology and chemistry lab tests, which will be measured against standard laboratory acceptable ranges for premature infants.

SECONDARY OUTCOMES:
Efficacy endpoint: Time to pneumatosis resolution | From date of NEC diagnosis until resolved, up to 10 days
  Pneumatosis is considered resolved when no longer observed on abdominal x-ray
Efficacy endpoint: Time to full enteral nutrition assessment | From date of completion of antibiotics and/or IP treatment until full feeding tolerance reached, 3-5 days
  Defined as no longer receiving total parenteral nutrition (TPN)
Efficacy endpoint: Incidence of abdominal surgical intervention | Assessed from Day 1/Baseline visit through 24 months of age
  Abdominal surgical intervention defined as laparotomy, including drain placement
Efficacy endpoint: Change in Neonatal Sequential Organ Failure Assessment (nSOFA) score | From Randomization/Day 1 through Day 10 of treatment period (10 days).
  nSOFA score is a neonatal sequential organ failure assessment of three organ systems: respiratory score criteria (range: 0-8); cardiovascular score criteria (range: 0-4); and Hematologic score criteria (range: 0-3) with a total score range: 0 (best) to 15 (worst)

OTHER OUTCOMES:
Exploratory endpoint: All cause mortality | From Day1/Baseline through 24 months of age
  Assessment of all deaths that occurred during the study
Exploratory endpoint: Length of stay in the NICU | From Day1/Baseline until date released from NICU - through 24 months of age
  Defined as total number of days from Day1/Baseline until date released from NICU
Exploratory endpoint: Change in weight over time | From Day1/Baseline through 24 months of age
  Weight will be measured in grams (g)
Exploratory endpoint: Change in length over time | From Day1/Baseline through 24 months of age
  Length will be measured in centimeters (cm)
Exploratory endpoint: Change in head circumference over time | From Day1/Baseline through 24 months of age
  Circumference will be measured in centimeters (cm) and will be used to ensure normal head growth.
Exploratory endpoint: Number of significant apnea events/day over time | From Day1/Baseline through 1 month follow-up visit - up to 2 months
  Significant apnea: any apnea for greater than 20 seconds
Exploratory endpoint: Number of significant bradycardia events/day over time | From Day1/Baseline through 1 month follow-up visit - up to 2 months
  Significant bradycardia: any bradycardia heart rate < 70BPM for > 6 seconds
Exploratory endpoint: Number of significant temperature instability events/day over time | From Day1/Baseline through 1 month follow-up visit - up to 2 months
  Significant temperature instability event: temperature < 36.5C or > 37.5C outside neutral/thermal environment or requires a change in isolette temperature outside of standard protocol
Exploratory endpoint: Time to return to normal bowel sounds | From date of NEC diagnosis until resolved, up to 10 days
  Defined as are typically soft and gurgling, indicating pneumatosis resolution and no feeding intolerance, no bowel obstruction or perforation.
Exploratory endpoint: Change in serum C-reactive protein (CRP) | To be assessed on Day2 and Day8 during treatment period; and 2 weeks and 1 month post treatment
  Included as part of labs being assessed per standard of care treatment
Exploratory endpoint: Time to return to normal serum platelet count levels | To be assessed on Day2 and Day8 during treatment period; and 2 weeks and 1 month post treatment
  Included as part of labs being assessed per standard of care treatment
Exploratory endpoint: Incidence of intestinal or colonic strictures | From Day1/Baseline through Day28/1 month post treatment follow up visit
  Measured by fluoroscopic study (barium enema or upper gastrointestinal scope); only conducted if infant had symptoms indicating partial bowel obstruction (e.g., feeding intolerance, abdominal distension, bilious emesis).
Exploratory endpoint: Incidence of sepsis | From Day1/Baseline through Day 28/1 month post treatment follow up visit
  Defined as presence of a pathogenic bacteria in blood culture or two positive blood cultures
Exploratory endpoint: Incidence of retinopathy | From Day1/Baseline until resolved - through 24 months of age
  To be monitored while in NICU
Exploratory endpoint: Incidence of bronchopulmonary dysplasia (BPD) | At 36 weeks of age and at discharge from NICU - up to 6 months
  To be identified at 36 weeks CGA and at discharge from NICU
Exploratory endpoint: Incidence of pulmonary hypertension (PH) | At 36 weeks of age and at discharge from NICU - up to 6 months
  To be identified at 36 weeks CGA and at discharge from NICU
Exploratory endpoint: Incidence of periventricular leukomalacia | From Day 1 post treatment follow up visit through 24 months of age
  To be measured via any form of imaging and noted if any symptoms observed

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Orlando Health, Inc. Winnie Palmer Hospital for Women and Babies, Orlando, Florida
  - BayCare Health System-St. Joseph's Women's Hospital, Tampa, Florida
  - NorthShore University-Evanston Hospital, Evanston, Illinois
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Oklahoma Children's Hospital, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center Magee Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No